CLINICAL TRIAL: NCT07158359
Title: Chewing Gum as a Therapeutic Intervention for the Management of Hypersalivation : a Pilot Study L'Utilisation du Chewing-gum Dans la Prise en Charge de l'hypersialorrhée : Une étude Pilote
Brief Title: Chewing Gum as a Therapeutic Intervention for the Management of Hypersalivation
Acronym: Chew Daily
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Cadillac (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-A00525-44; IDRCB (Other: ANSM)
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Hypersialorrhea (Excessive Salivation); Psychiatric Disorders
Keywords: Rehabilitation; occupational therapy; pilot study; chewing gum mastication; non-pharmacological treatment
MeSH Terms: conditions — Sialorrhea; Mental Disorders

STUDY DESIGN:
Intervention Model Description: This study falls within the field of Research Involving Human Participants. It is classified as Category 2: interventional research involving minimal risk. The study is designed as a prospective, longitudinal investigation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group assigned to a swallowing rehabilitation program involving chewing gum mastication (Experimental): Each participant will receive a rehabilitation session (including chewing gum mastication) three times per week over a four-week period. Each session will last 15 minutes (i.e., 10 minutes of mastication followed by a 5-minute waiting period prior to reassessment). The 10-minute mastication period was determined based on clinical feedback from patients regarding this practice. Rehabilitation sessions will always take place at least 30 minutes after meals.
  During each mastication session, the participant will be observed in a quiet room, with a comic book available for distraction. Hypersialorrhea will be assessed three times per session using the DSFS scale: immediately before chewing gum mastication, at the end of the mastication period, and 5 minutes thereafter.
  The rehabilitation program will run over four weeks, from Monday to Friday, corresponding to 12 non-consecutive days. The four-week duration was chosen in accordance with standard occupational therapy clinical practice. In
  Interventions: Behavioral: chewing gum mastication
- Control group (No Intervention): For the control group, which will not receive any rehabilitation, the same schedule will be followed. Each participant will be seen three times per week for 15 minutes. During these observation sessions (no intervention, absence of any rehabilitation), hypersialorrhea will be assessed three times using the DSFS scale: immediately before, at the end of the 10-minute period, and 5 minutes thereafter.
  During these observation sessions, participants will be placed in a quiet room with a comic book available for distraction. The observation period will span four weeks, corresponding to 12 non-consecutive days. In parallel, the healthcare team will be asked to respond three times per week to a single adherence-related question during the scheduled sessions.

INTERVENTIONS:
Behavioral: chewing gum mastication — chewing gum mastication
  Arms: Experimental group assigned to a swallowing rehabilitation program involving chewing gum mastication

SUMMARY:
Psychiatric disorders often require specific treatments, usually involving medications called psychotropic drugs. While effective, these medications can cause significant side effects. One of the most common is hypersalivation (excess saliva), which can make swallowing difficult and be very uncomfortable in daily life.

Current medication-based solutions are often not very effective and may cause additional side effects. For this reason, we are exploring a different approach: using chewing gum as a form of rehabilitation.

The goal of this study is to determine whether chewing gum can help reduce excessive saliva. To do this, we will compare two groups: one that will follow a swallowing rehabilitation program including chewing gum, and another that will not.

We hope this simple, non-drug-based approach will improve the management of hypersalivation. More broadly, this research aims to highlight innovative and accessible solutions in psychiatry, showing that alternative strategies-sometimes very simple ones-can also be effective.

DETAILED DESCRIPTION:
Introduction Psychiatric disorders necessitate highly specific therapeutic approaches. Psychotropic medications, which are frequently prescribed in these settings, are well known for their substantial burden of adverse drug reactions. Among these, hypersialorrhea (excessive salivation) is a particularly common and disabling side effect, often associated with swallowing disturbances. Current pharmacological alternatives proposed to address this condition remain of limited efficacy and may themselves induce additional adverse effects. In light of these limitations, a rehabilitative, non-pharmacological intervention such as chewing gum mastication may represent a promising strategy.

Objective The primary objective of this pilot study is to assess the effect of chewing gum mastication on hypersialorrhea in patients receiving psychotropic medications.

Methods A randomized controlled trial will be conducted, comparing two groups: an experimental group undergoing a swallowing rehabilitation program incorporating chewing gum mastication, and a control group receiving no chewing-gum-based intervention.

Expected Results This study is expected to provide preliminary evidence supporting the clinical utility of chewing gum mastication as a non-pharmacological approach for the management of hypersialorrhea. Beyond its direct clinical implications, the study aims to promote awareness of innovative, unconventional, yet potentially effective therapeutic strategies in psychiatry, thereby fostering further research in this field.

Keywords Rehabilitation; occupational therapy; psychiatry; pilot study; chewing gum mastication; clinical management; non-pharmacological treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years.
* Hospitalized at Cadillac Hospital, either in full inpatient care or at the rehabilitation facility, excluding the UHSA.
* Experiencing iatrogenic hypersalivation induced by psychotropic medications.
* Salivary flow causing functional impairment for the patient, or observed by family members or healthcare providers.
* With or without pharmacological management of hypersalivation.
* Individuals under legal protective measures may be included.
* Provided written informed consent prior to participation.

Exclusion Criteria:

* Anatomical/morphological anomaly affecting mastication/swallowing
* Swallowing disorder of organic etiology (e.g., neurological deficit due to stroke, neurodegenerative disease, oropharyngeal surgery, etc.)
* Known risk of aspiration with liquids
* Patient refusal of chewing gum or inability to obtain consent (e.g., non-communicative patients)
* Oral/dental condition preventing mastication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Salivary flow measured using the Drooling Severity and Frequency Scale (DSFS) in relation to chewing gum mastication | 4 weeks

SECONDARY OUTCOMES:
Quality of life, evaluated with the Clinical Global Impression (CGI), was assessed pre- and post-experimental phase | 4 weeks
Patient adherence to medication will be assessed weekly by the healthcare team using a single dichotomous question: "Did the patient demonstrate opposition to taking their medication related to hypersalivation?" | 4 weeks
Use of pharmacological agents associated with adverse effects will be monitored through prescription tracking. | 4 weeks
Tolerance and safety of chewing gum as a therapeutic intervention will be evaluated by the investigative team at each session using two dichotomous questions: "Did you observe any tolerance or safety issues during chewing gum mastication in this session? | 4 weeks

IPD SHARING:
Plan to Share IPD: No